CLINICAL TRIAL: NCT01430416
Title: A Phase 1 Study of AEB071, an Oral Protein Kinase C Inhibitor, in Patients With Metastatic Uveal Melanoma
Brief Title: Safety and Efficacy of AEB071 in Metastatic Uveal Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COEB071X2102; 2011-002535-25 (EudraCT Number)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-05

CONDITIONS: Uveal Melanoma
Keywords: Uveal melanoma; phase 1; AEB071; Metastatic
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — sotrastaurin

ARMS (1):
- AEB071 (Experimental)
  Interventions: Drug: AEB071

INTERVENTIONS:
Drug: AEB071

SUMMARY:
This study has two parts, dose escalation and dose expansion. For dose escalation, the primary objective is to estimate the maximum tolerated dose (MTD) of AEB071 in patients with uveal melanoma. For dose expansion, the primary objective is to characterize the safety and tolerability of the MTD of AEB071 in patients with uveal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Uveal melanoma with biopsy proven metastatic disease
* Males and females ≥ 18 years of age
* Consent to biopsy of tumor
* Measurable disease according to RECIST version 1.1
* WHO performance status of ≤ 1

Exclusion Criteria:

* Patients with abnormal laboratory values as defined by the protocol
* Patients who are receiving treatment with strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) that cannot be discontinued prior to study entry
* Patients with impaired cardiac function or clinically significant cardiac diseases as defined by the protocol
* Patients with another malignancy that was treated within the last three years with the exceptions of localized basal cell carcinoma and cervical carcinoma
* Patients with impairment of gastrointestinal function or disease
* Patients with severe systemic infections
* Patients who are known to be HIV positive and/or have active hepatitis B or C infection
* Time since last therapy for treatment of underlying malignancy:

  * Cytotoxic chemotherapy: ≤ duration of the most recent cycle of the previous regimen (a minimum of 2 weeks for all)
  * Nitrosurea: ≤ 6 weeks
  * Biologic therapy: ≤ 4 weeks
  * ≤ 5 x PK half-life of a small molecule therapeutic not otherwise defined above
* Patients having undergone major surgery less than 4 weeks prior to enrollment or have not fully recovered from prior surgery
* Women of child-bearing potential unless they are using highly effective methods of contraception during the dosing and for at least 36 hours after last dose. Highly effective contraception as defined in the protocol.
* Patients with primary central nervous system tumors or brain metastases.
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-12-20 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicity during cycle 1 (28 days) - Dose Escalation | cycle 1 (28 days)
Number of participants reporting serious adverse events and adverse events - Dose Expansion | Baseline, every 28 days

SECONDARY OUTCOMES:
Overall response rate (Complete Response (CR) + Partial Response(PR)) to AEB071 using RECIST version 1.1 | Baseline, 12 months
Progression free survival and time to progression using RECIST version 1.1 | Baseline, 12 months
Number of patients reporting serious adverse events and adverse events | Baseline, 12 months
AEB071/AEE800 pharmacokinetic parameters including Cmax, tmax, AUCτ, Ctrough, CL/F, and RA | First 7 months of treatment period
Gα genotype in tumor specimens | Baseline, 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - Dana Farber Cancer Institute DFCI - Brookline, Boston, Massachusetts
  - Memorial Sloan Kettering MSKCC 4, New York, New York
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- See also: Results for COEB071X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17658